CLINICAL TRIAL: NCT05566470
Title: Assessment of Central Neuromuscular Dysfunction, Shoulder Physical Functionality and Psychological Factors in Individuals Undergoing Rotator Cuff Surgery
Brief Title: Central Neuromuscular Dysfunction, Functionality, Psychological Status and Rotator Cuff Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gizem Irem KINIKLI, Gizem İrem Kınıklı, Assoc., Prof., PT, Hacettepe University
Other Study IDs: GO 22/643
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Tears
Keywords: Transcranial magnetic stimulation; Rotator Cuff Tear; Functionality; Psychological Resilience; Depression, anxiety, stress; Central Neuromuscular Function
MeSH Terms: conditions — Rotator Cuff Injuries; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: 1. Healty adults aged between 30-65 years old who do not have any pathology related to the shoulder joint and have not undergone surgery and being a volunteer to participate in the study.
  Interventions: Diagnostic Test: Assessment of Central Neuromuscular Dysfunction, Shoulder Physical Functionality and Psychological Factors
- Patient Group: 1. Individuals between 30-65 years old who have been diagnosed with massive rotator cuff tear,
  2. At least 6 months have passed after the surgery,
  3. In the last 6 months, patients have not undergone shoulder surgery except for rotator cuff tear surgery,
  4. Arthroscopic surgical method was performed by Prof. Dr. Gazi Huri,
  5. The absence of another lesion involving the shoulder joint, such as SLAP (Superior Labrum Anterior Posterior), recurrent shoulder dislocation, arthroplasty, except for massive complete tear in the patient will be included in the study
  Interventions: Diagnostic Test: Assessment of Central Neuromuscular Dysfunction, Shoulder Physical Functionality and Psychological Factors

INTERVENTIONS:
Diagnostic Test: Assessment of Central Neuromuscular Dysfunction, Shoulder Physical Functionality and Psychological Factors — Each of the 2 groups will be evaluated in terms of functional level and psychological factors; American Shoulder and Elbow Surgeons evaluation form (ASES), Connor-Davidson Psychological Resilience Scale (CDPRS) and the Depression, Anxiety, Stress-21 Scale (DASS-21) will be used to evaluate these factors. Furthermore, the corticospinal excitability of the deltoid muscle will be assessed with Transcranial Magnetic Stimulation (TMS). Both deltoid muscles of the patient will be evaluated by saving motor evoked potentials signals that respond to TMS, and motor excitability will be compared between the affected arm and the unaffected arm. In addition, the control group will also be assessed in terms of functional level and psychological factors with TMS, ASES, DASS-21 and CPDRS.

SUMMARY:
Considering the fact that The problems experienced by the patients are not only physiological but also psychological and social. Unfortunately, there is no sufficient study focus on all these concepts.

Generally, studies focus on only physiological dimensions such as functional level, muscle strength and pain. The aim of this study, in addition to assessment methods commonly used for functional level, muscle strength and pain, is to evaluate central neuromuscular function on individuals who have undergone rotator cuff tear surgery with transcranial magnetic stimulation. Furthermore, psychological resilience, which is considered as a positive psychological trait, will also be evaluated. Until now, only one study has evaluated the role of psychological resilience in the postoperative process of rotator cuff surgery. This study has shown that the correlation between functionality and psychological resilience. As a result of our study, the influence of resiliency on postoperative outcomes following rotator cuff surgery will be determined and central neuromuscular function, shoulder functional level, and psychological resilience changes will be revealed in physiological and psychological concepts.

Furthermore, this study may show that psychological resilience has a potential role on predicting functional level and pain.

It is planned that the results obtained will guide the postoperative rehabilitation of rotator cuff surgery for further studies on multidimensional perspectives.

DETAILED DESCRIPTION:
The problems experienced by the patients are not only physiological but also psychological and social. Unfortunately, there is no sufficient study focus on all these concepts.

For all these reasons, it is seen that in order to offer an individualized rehabilitation program to patients, it is needed to add psychological evaluation methods that can directly affect the results of treatment as well as physical and objective evaluations during the evaluation phase.

As a physical evaluation method, the cortico-spinal excitability of the deltoid muscle will be evaluated with the Transcranial Magnetic Stimulation (TMS) to determine the effects of rotator cuff tears on the central neuromuscular function of the upper extremity muscles in patients who have undergone rotator cuff tear surgery.

Superficial electromyography (EMG) studies have shown that central neuromuscular dysfunction of deltoid muscle in chronic rotator cuff tears is associated with activation of adjacent shoulder muscles. Until now, only one study has evaluated the central neuromuscular function of deltoid muscle with Transcranial Magnetic Stimulation (TMS).

Transcranial Magnetic Stimulation (TMS) is a non-invasive evaluation method in which magnetic fields are used to stimulate neural structures such as cerebral cortex, spinal roots, cranial and spinal neurons and the responses resulting from these stimulations are recorded with EMG device One of the main symptoms of patients with Rotator Cuff Tear is pain. According to John et al. and Martinez et al., psychological resilience is an important factor during coping with pain. Higher phological resilience has been associated with less pain intensity, less pain-related limitations, more social support, and more pain self-efficacy. The American Psychological Association (2014) defines resilience as "the process of adapting well in the face of adversity, trauma, tragedy, threats or even significant sources of stress." Studies has shown that resilience has a potential role for patient recovery. Until now, only one study has evaluated the role of psychological resilience in the postoperative process of rotator cuff surgery.

Therefore, the main purpose of this study is to investigate the relationship of central neuromuscular function of deltoid muscle with functional level and psychological factors.

The psychological factors that will be evaluated are depression, anxiety, stress and psychological resilience. The effect of these psychological factors on functional level will also be examined.

Considering that psychological resilience is also associated with social participation, higher psychological resilience allows patients to receive better social support during the rehabilitation process and communicate more effectively with their environment.

As a result of our study, the influence of resiliency on postoperative outcomes following rotator cuff surgery will be determined and central neuromuscular function, shoulder functional level, and psychological resilience changes will be revealed in physiological and psychological concepts.

Furthermore, this study may show that psychological resilience has a potential role on predicting functional level and pain.

It is planned that the results obtained will guide the postoperative rehabilitation of rotator cuff surgery for further studies on multidimensional perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Patient Group:

  1. Volunteer to participate in the study,
  2. Be between the ages of 30 and 65,
  3. Individuals who have been diagnosed with massive rotator cuff tear and the who have undergone rotator cuff tear surgery,
  4. At least 6 months have passed after the surgery,
  5. In the last 6 months, patients have not undergone shoulder surgery except for rotator cuff tear surgery,
  6. Arthroscopic surgical method was performed by Prof. Dr. Gazi Huri,
  7. The absence of another lesion involving the shoulder joint, such as SLAP (Superior Labrum Anterior Posterior), recurrent shoulder dislocation, arthroplasty, except for massive complete tear in the patient will be included in the study.
* Inclusion Criteria for Control Group :

  1. Demographic characteristics (age and gender) similar to the study group,
  2. Not having any diagnosis related to the shoulder joint.

Exclusion Criteria:

1. Having any additional pathology (SLAP (Superior Labrum Anterior Posterior), recurrent shoulder dislocation, arthroplasty etc.) concerning the shoulder joint,
2. Having a history of surgery involving the shoulder,
3. Having a neuromuscular and/or metabolic disease,
4. Presence of active infection
5. Other coexisting neuromuscular and musculoskeletal pathologies,
6. To have been diagnosed with bilateral RMY,
7. Metal implants in the head and neck,
8. Being pregnant,
9. Those who use drugs that can change cortical excitability,
10. Being a cancer patient,
11. Individuals with cognitive and psychiatric disorders will not be included in this study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 17 individuals, male and female, between the ages of 30-65 who have undergone rotator cuff tear surgery, will be included in the study. 17 healthy individuals from the close circle of the researchers reached by snowball method will be included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Transcranial Magnetic Stimulation (TMS) | 1 day
  Transcranial Magnetic Stimulation (TMS) will be used to evaluate corticomotor excitability. TMS is a non-invasive evaluation method in which magnetic fields are used to stimulate neural structures such as cerebral cortex, spinal roots, cranial and spinal neurons and the responses resulting from these stimulations are recorded with electromyography (EMG) device and is used for prognostic and evaluation purposes.
The American Shoulder and Elbow Surgeons Score (ASES) | 1 day
  ASES Standardized Shoulder Assessment form was used to evaluate patient-rated shoulder pain and function. ASES consists of two parts in which therapists evaluate patients and patients evaluate themselves. The questionnaire includes questions about patients' pain and activities of daily living. Evaluation is made over 100 points. 0 is the minimum score, 100 is the maximum points. Higher scores indicate a better functional level.
Connor-Davidson Psychological Resilience Scale (CDPRS) | 1 day
  It was developed to measure psychological resilience. The answers to the scale are sorted as 0: not correct at all, 1: rarely correct, 2: sometimes correct, 3: often correct, 4: almost always correct. Each question is scored between 0 and 4 points. There are 3 sub-dimensions of the scale. Perseverance and personal competence, tolerance to negative phenomena and spiritual inclination are the main headings of the 3 sub-dimensions. The highest score to be obtained from the first sub-dimension, perseverance and personal competence, is 60, the highest score that can be obtained from tolerance to negative phenomena, which is the second sub-dimension, is 24, and the highest score to be obtained from the third sub-dimension, spiritual tendency, is 16. In conclusion, evaluation is made over 100 points. 0 is the minimum score, 100 is the maximum points. Higher scores indicate a better resilience status.
Depression, Anxiety, Stress-21 Scale (DASS-21) | 1 day
  The scale is used to measure the symptoms of depression, anxiety and stress both in the clinical sample and in the normal sample.
  In this measurement tool, the 0-7 score range is normal depression, the 0-7 point range is normal anxiety, and the 0-14 point range is normal stress indicator. There are 7 questions to measure each of the dimensions of depression, stress and anxiety. On the scale, 0 is scored as "never", 1 as "sometimes", 2 as "quite often", and 3 as "always".
  The fact that the individual receives 5 points and above from the depression sub-dimension, 4 points and above from anxiety, and 8 points and above from stress shows that the symptoms are not normal.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Sena Yarımkaya, BSc., Principal Investigator — Atılım University; Gizem İrem Kınıklı, Assoc. Prof., Study Chair — Hacettepe University
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Porter A, Hill MA, Harm R, Greiwe RM. Resiliency influences postoperative outcomes following rotator cuff repair. J Shoulder Elbow Surg. 2021 May;30(5):1181-1185. doi: 10.1016/j.jse.2020.08.024. Epub 2020 Sep 9. PMID 32919049
- [Background] Berth A, Pap G, Awiszus F, Neumann W. Central motor deficits of the deltoid muscle in patients with chronic rotator cuff tears. Acta Chir Orthop Traumatol Cech. 2009 Dec;76(6):456-61. PMID 20067692
- [Background] Nollet H, Van Ham L, Deprez P, Vanderstraeten G. Transcranial magnetic stimulation: review of the technique, basic principles and applications. Vet J. 2003 Jul;166(1):28-42. doi: 10.1016/s1090-0233(03)00025-x. PMID 12788015
- [Background] Hassett AL, Finan PH. The Role of Resilience in the Clinical Management of Chronic Pain. Curr Pain Headache Rep. 2016 Jun;20(6):39. doi: 10.1007/s11916-016-0567-7. PMID 27115770